CLINICAL TRIAL: NCT00003097
Title: Skin Cancer Prophylaxis by Low-Fat Dietary Intervention
Brief Title: Low Fat Diet to Prevent Disease Progression in Patients With Skin Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000065820; BCM-H-109; NCI-P97-0105
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-10

CONDITIONS: Non-Melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell

INTERVENTIONS:
Other: preventative dietary intervention

SUMMARY:
RATIONALE: A low-fat, balanced diet may prevent disease progression in patients with nonmelanomatous skin cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of a low-fat, balanced diet to prevent disease progression in patients with nonmelanomatous skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether intervention with a low-fat balanced diet will prolong the disease-free survival time in patients presenting with nonmelanomatous skin cancer and having a history of not more than two previous skin cancers. II. Assess the effect of this intervention on numbers of tumors during the two year follow-up period. III. Determine the incidence of new skin cancer in the control, nonintervention population.

OUTLINE: This is a randomized study. Patients are randomized into the Dietary Intervention or Nonintervention groups. The control group has initial and follow up assessment of eating habits. The dietary intervention group also has initial and follow up assessment of eating habits that have been changed to reduce fat intake to one-half of the amount in the average American diet with a subsequent increase of carbohydrates to compensate for total caloric intake. Both groups have assessment of clinical status of skin cancer at 4 month intervals for 24 months. Patients are followed for two years.

PROJECTED ACCRUAL: Approximately 175 patients will be accrued in the first 3 years of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed basal cell carcinoma or squamous cell carcinoma of the skin No more than two prior skin carcinomas Must not have genetic predisposition to skin cancer (i.e., xeroderma pigmentosum, basal cell nevous syndrome)

PATIENT CHARACTERISTICS: Age: 15 and over Race: Caucasian Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No therapeutic diet that requires fat intake greater than 20% of total calories No untreated systemic malignancy No history of arsenic ingestion Not diabetic

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent systemic steroids Radiotherapy: No prior x-ray therapy for acne No prior/concurrent ultraviolet light (PUVA or UVB) therapy for psoriasis Surgery: Not specified Other: No concurrent megavitamin or mineral supplementation At least 5 years since treatment with antimetabolites, folic acid inhibitors, alkalating agents, etc.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 1989-04

CONTACTS AND LOCATIONS:
Overall Officials: Homer Black, PhD, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Black HS, Jaax S: Low-Fat Dietary Guide to Aid in the Management of Skin Cancer. Houston, TX: 1999.
- [Background] Black HS. Influence of dietary factors on actinically-induced skin cancer. Mutat Res. 1998 Nov 9;422(1):185-90. doi: 10.1016/s0027-5107(98)00191-2. PMID 9920444
- [Background] Black HS: Diet and skin cancer. In: Heber D, Blackburn GL, Go VL: Nutritional Oncology. San Diego, CA: Academic Press, 1999, pp. 405-419.
- [Background] Jaax S, Scott LW, Wolf JE Jr, Thornby JI, Black HS. General guidelines for a low-fat diet effective in the management and prevention of nonmelanoma skin cancer. Nutr Cancer. 1997;27(2):150-6. doi: 10.1080/01635589709514517. PMID 9121942
- [Result] Black HS, Wolf JE: Protective influence of a low-fat diet on non-melanoma skin cancer. Dermatologic Therapy: Phototherapy and Photoprotective Therapy 4: 100-105, 1997.
- [Result] Black HS, Wolf JE: A low-fat diet can reduce skin cancer risk. Primary Care and Cancer 15: 12-13, 1996.
- [Result] Black HS: Low-fat diet impedes the development of actinic keratosis. Biomedical Pharmacotherapy 49: 46-47, 1995.
- [Result] Black HS, Thornby JI, Wolf JE Jr, Goldberg LH, Herd JA, Rosen T, Bruce S, Tschen JA, Scott LW, Jaax S, et al. Evidence that a low-fat diet reduces the occurrence of non-melanoma skin cancer. Int J Cancer. 1995 Jul 17;62(2):165-9. doi: 10.1002/ijc.2910620210. PMID 7622291
- [Result] Black HS, Wolk JE Jr: A low-fat diet can reduce skin cancer risk. Skin Cancer Foundation Journal 13: 37/98, 1995.
- [Result] Black HS, Herd JA, Goldberg LH, Wolf JE Jr, Thornby JI, Rosen T, Bruce S, Tschen JA, Foreyt JP, Scott LW, et al. Effect of a low-fat diet on the incidence of actinic keratosis. N Engl J Med. 1994 May 5;330(18):1272-5. doi: 10.1056/NEJM199405053301804. PMID 8145782